CLINICAL TRIAL: NCT04351490
Title: Impact of Zinc and Vitamin D3 Supplementation on the Survival of Institutionalized Aged Patients Infected With COVID-19
Brief Title: Impact of Zinc and Vitamin D3 Supplementation on the Survival of Aged Patients Infected With COVID-19
Acronym: ZnD3-CoVici
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: change study design and funding
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020_30; 2020-A00873-36 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2020-04

CONDITIONS: SARS-CoV 2
Keywords: Survival; Covid-19; Aged subjects; Zinc; 25-OH cholecalciferol
MeSH Terms: conditions — COVID-19 | interventions — gluconic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group supplementation (Experimental)
  Interventions: Dietary Supplement: Zinc gluconate; Dietary Supplement: 25-OH cholecalciferol
- Group usual treatment (No Intervention)

INTERVENTIONS:
Dietary Supplement: Zinc gluconate — Zinc gluconate capsule 15 mg x 2 per day during 2 months
  Arms: Group supplementation
Dietary Supplement: 25-OH cholecalciferol — 25-OH cholecalciferol drinkable solution 10 drops (2000 IU) per day during 2 months
  Arms: Group supplementation

SUMMARY:
Mortality from Covid-19 increases with age, reaching 14.8% from the age of 80. The severity of the infection is linked to the acute respiratory distress syndrome (ARDS) which requires intensive care. ARDS is the consequence of the reactional inflammatory storm that damages the lungs.

Aged subjects are particularly prone to zinc and vitamin D deficiency. These two micronutrients are able to modulate the immune response by reducing the inflammatory storm.

The hypothesis is that supplementation with zinc and vitamin D would reduce the inflammatory reaction which worsens ARDS and leads to the death of subjects infected with Covid-19.

ELIGIBILITY:
Inclusion Criteria:

* Institutionalized

Exclusion Criteria:

* Life expectancy < 1 month independently of Covid-19 infection (overall subjects)
* Known hypercalcemia
* History of renal lithiasis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Survival rate in asymptomatic subjects at inclusion | Two months after inclusion

SECONDARY OUTCOMES:
Survival rate in symptomatic subjects at inclusion | Two months after inclusion
Survival rate in overall subjects | Two months after inclusion
  symptomatic subjects and asymptomatic subjects
Cumulative incidence of Covid-19 infection in asymptomatic subjects at inclusion | Within two months after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: David SEGUY, MD,PhD, Principal Investigator — University Hospital, Lille

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shakoor H, Feehan J, Al Dhaheri AS, Cheikh Ismail L, Ali HI, Alhebshi SH, Apostolopoulos V, Stojanovska L. Role of vitamin D supplementation in aging patients with COVID-19. Maturitas. 2021 Oct;152:63-65. doi: 10.1016/j.maturitas.2021.03.006. Epub 2021 Mar 16. No abstract available. PMID 33757717